CLINICAL TRIAL: NCT06445660
Title: The Feasibility of a Radiological Score Based on Quantified Analysis of Computed Tomography Signs for Recognizing Salvageable Bowel in Acute Mesenteric Ischemia: A Retrospective Analysis of Prospective Study
Brief Title: The Feasibility of a Radiological Score Based on CT Signs for Recognizing Salvageable Bowel in Acute Mesenteric Ischemia
Acronym: AMESIradiol
Status: Recruiting | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Annika Reintam Blaser, associate professor, University of Tartu
Other Study IDs: 03.01.2024
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: Patients included in the AMESI study as suspected AMI
- AMI patients with salvageable bowel: Patients included in the AMESI study with confirmed AMI, who did not undergo bowel resection
  Patients with one of the following:
  1. treated endovascularly and did not undergo bowel resection secondarily
  2. received surgical revascularization without bowel resection (initial or secondary)
  3. received explorative laparoscopy or laparotomy without the need for bowel resection (initially or secondarily)
  4. received conservative treatment without the need for secondary bowel resection
- AMI patients with non-salvageable bowel: Patients included in the AMESI study with confirmed AMI who (one of the following):
  1. underwent bowel resection initially
  2. underwent bowel resection secondarily
  3. did not undergo bowel resection because non-salvageable bowel
  4. were changed to palliation due to the progression of ischaemia after any initial treatment with curative intention (including endovascular and conservative)

SUMMARY:
Computed tomography (CT) is the standard modality for scanning patients with critical acute abdominal conditions, including suspected acute mesenteric ischemia (AMI). CT imaging can potentially differentiate between reversible and irreversible ischaemic damage of the bowel. This moment is pivotal in selecting the treatment strategy for AMI - in the absence of irreversible damage; reperfusion therapy can preserve intestinal viability, thereby avoiding the need for bowel resection. The present study tests the hypothesis that combining several symptoms may enhance the diagnostic performance of CT scanning in detecting salvageable bowel in patients with AMI. This study is an ancillary component of the AMESI study (Clinical Trials: NCT05218863) - a prospective, multicentre observational study aimed at identifying the incidence and describing the outcomes of acute mesenteric ischemia (AMI) in adult hospitalized patients. The ultimate purpose of the present study is to create a computed tomography-based radiological score for the assessment of bowel viability in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

* Participant in AMESI study
* confirmed or suspected acute mesenteric ischaemia
* CT scan of the entire abdominal cavity / full body using intravenous contrast media is available

Exclusion Criteria:

* Scans without the use of an intravenous contrast media or those covering only a partial area of the abdomen will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a substudy of the AMESI study - "Incidence, Diagnosis, Management, and Outcome of Acute Mesenteric Ischaemia: A Prospective, Multicentre Observational Study." (Clinical Trials: NCT05218863) As of the end of August 2023, a total of 705 patients from 32 study sites worldwide have been enrolled, with 418 of them having confirmed cases of AMI. For patients with confirmed AMI, comprehensive data collection concerning diagnostics, management, and long-term outcomes has been completed
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency rate | up to one month
  Frequency rate of common radiological signs in AMI patients with and without salvageable bowel.

SECONDARY OUTCOMES:
Performance of the radiological score | up to one month
  Performance of the radiological score in patients with different types of AMI.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Starkopf, Study Chair — University of Tartu, Department of Anaesthesiology and Intensive Care
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT06445660/Prot_000.pdf